CLINICAL TRIAL: NCT06522581
Title: Role of Citicoline in Treatment of Neonates With Hypoxic Ischemic Encephalopathy
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Armed Forces Hospital, Pakistan (Other)
Responsible Party: Principal Investigator, arshad khushdil, Doctor, Armed Forces Hospital, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Citicoline for HIE
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Hypoxic Ischemic Encephalopathy of Newborn

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- neonates with HIE receiving citicoline (Experimental): this arm will include neonates suffering from hypoxic ischemic encephalopathy and who will be given injection citicoline
  Interventions: Drug: Citicoline Sodium
- neonates with HIE receiving placebo (Placebo Comparator): this arm will include neonates who will be suffering from HIE but will recieve rotuine care in NICU but will not receive injection citicoline
  Interventions: Drug: Citicoline Sodium

INTERVENTIONS:
Drug: Citicoline Sodium — one group of neonates with confirmed HIE grade II and III will receive injection citicoline through IV route within 06 hours of birth
  Other Names: placebo

SUMMARY:
Hypoxic ischemic encephalopathy is an acute or subacute brain injury, due to asphyxia in neonates, leading to mortality and long-term morbidity. Its prevalence varies across regions, with developed countries reporting rates of 1.5 per 1000 live births, while developing nations experience a wider range from 2.3 to 26.5 per 1000 live births.

Infants afflicted with moderate HIE face a 10% risk of mortality, with surviving individuals encountering a 30% chance of developing disabilities. The prognosis is graver for severe HIE, with a mortality risk of 60%, and nearly all survivors experiencing some form of disability.

DETAILED DESCRIPTION:
A number of treatment modalities are available but are not clinically effective due to inefficacy and undesirable side effects. Despite therapeutic hypothermia being the sole effective neuroprotector to date, its applicability is limited in certain scenarios, such as gestational age below 36 weeks, birth weight under 2000 g, and initiation beyond 6 hours of age. Therefore, there is a critical need to explore alternative, safe, effective, and accessible neuroprotective therapies, particularly in developing nations.

Citicoline, cytidine 5-diphosphocholine, is an exogenous substance and a product of rate limiting step of phosphatidyl choline synthesis. It has rapid absorption through enteral route where it breaks into cytidine and choline. Citicoline is a favorable recently developed neuroprotector in HIE as it helps to regenerate neuronal cells by inhibiting different steps of ischemic cascade like inhibiting glutamate built up and ROS synthesis increasing dopamine and acetylcholine neurotransmitters, regenerating injured cell membrane and increasing brain plasticity and repair.

In this study, effects of citicoline as a neuroprotector are evaluated in neonates with moderate and severe HIE.

ELIGIBILITY:
Inclusion Criteria:

1. all indoor newborn babies with HIE II and III
2. who have not received therapeutic hypothermia

Exclusion Criteria:

1. grade I HIE
2. Babies on TH
3. babies whose parents do not give consent for inclusion in study
4. babies with major congential malformations -

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
survival in newborn babies with HIE | one year after the start of study
  we will be evaluationg the efficacy of citicoline in newborns with HIE

CONTACTS AND LOCATIONS:
Overall Officials: arshad Khushdil, FCPS, Principal Investigator — PEMH
Locations (1):
- MH, Rawalpindi, Pakistan